CLINICAL TRIAL: NCT07248501
Title: Effects of Bulgarian Bag Exercise on Lower Limb Function, Posture and Balance Among School Going Children
Brief Title: Effects of Bulgarian Exercises on Lower Limb Function in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/FAREEHASALEEM
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Child, Only
Keywords: Bulgarian exercise, Postural awareness scale PAS-E

STUDY DESIGN:
Intervention Model Description: The objective of this study is to investigate the Effect of Bulgarian bag exercises on lower limb function, posture and balance among school going students. In this investigation, our study will include 379 participants girls and boys in our study. Non-Probability Convenient sampling will be used in this research. In this investigation, will collect data from Lahore primary school going girls and boys. The sample that will be included in our study will be 8 to 16 years of age, with both genders, Informed consent, Healthy children without any diagnosed physical or neurological impairments that could affect motor skills or agility. This study use following tools in our study Postural awareness scale PAS-E, Berg balance scale, The lower extremity functional scale.
Masking Description: Participants will get same treatment protocols and possible efforts will be put to mask the group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Group(Bulgarian Bag Exercise Program) (Experimental): The Bulgarian Bag exercises will be performed under the guidance of a trained physical therapist or instructor. Key exercises will include squats, lunges, deadlifts, and shoulder presses, all performed with the Bulgarian Bag to target lower body strength, balance, and coordination. Progressions (e.g., increasing repetitions or load) will be made gradually as participants adapt to the exercises.
  Interventions: Other: Bulgarian Bag Exercises

INTERVENTIONS:
Other: Bulgarian Bag Exercises — The Bulgarian Bag exercises will be performed under the guidance of a trained physical therapist or instructor. Key exercises will include squats, lunges, deadlifts, and shoulder presses, all performed with the Bulgarian Bag to target lower body strength, balance, and coordination.
  Progressions (e.g., increasing repetitions or load) will be made gradually as participants adapt to the exercises.

SUMMARY:
The objective of this study is to investigate the Effect of Bulgarian bag exercises on lower limb function, posture and balance among school going students. In this investigation, our study will include 379 participants girls and boys in our study. Non-Probability Convenient sampling will be used in this research. In this investigation, will collect data from Lahore primary school going girls and boys. The sample that will be included in our study will be 8 to 16 years of age, with both genders, Informed consent, Healthy children without any diagnosed physical or neurological impairments that could affect motor skills or agility. This study use following tools in our study Postural awareness scale PAS-E, Berg balance scale, The lower extremity functional scale.

DETAILED DESCRIPTION:
Bulgarian Training Bag is a training equipment used in strength training, Plyometrics, Weight training, aerobic exercise, and fitness in general. Bags are made of leather or synthetic leather and filled with sand; Weigh between 3 to 38 kg and have flexible handles to allow training of the upper and lower body, and to improve the prehensile strength. Instead, Leisure Physical Activity should be thought of as all physical activity behavior that emanates from an unconscious drive for movement. Regular participation in physical activity is important for overall health. It provides children with immediate social, mental and physical health benefits, such as reducing symptoms of depression, improving academic and cognitive performance, promoting healthy bone structure, skeletal health supporting muscle growth and the development of the body's vital organs, particularly the heart and lungs, improving health related fitness, muscular strength and, preventing children from becoming overweight.

The objective of this study is to investigate the Effect of Bulgarian bag exercises on lower limb function, posture and balance among school going students. In this investigation, our study will include 379 participants girls and boys in our study. Non-Probability Convenient sampling will be used in this research. In this investigation, will collect data from Lahore primary school going girls and boys. The sample that will be included in our study will be 8 to 16 years of age, with both genders, Informed consent, Healthy children without any diagnosed physical or neurological impairments that could affect motor skills or agility. This study use following tools in our study Postural awareness scale PAS-E, Berg balance scale, The lower extremity functional scale.

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform physical activities
* Participants must be between 8 to 18 years

Exclusion Criteria:

* Children with severe physical disabilities or medical conditions that limit participation in physical activities (e.g., cardiovascular or respiratory conditions).
* Children unable to comply with study requirements or follow instructions

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 345 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Postural Awareness Scale PAS-E | 11 weeks
  Body posture refers to the position of a person's body in space and the alignment of body parts in relationship to one another and to the environment at one point in time. Postural awareness is informed via receptors in joints, muscles, ligaments, and connective tissue, which is then integrated in the central nervous system. Importantly, postural awareness is influenced by mental processes, including attention, interpretation, and appraisal of bodily sensation, as well as by affect, emotions, and attitudes.
Pediatrics Berg Balance Scale | 11 weeks
  The Berg Balance Scale has proven to be a reliable and valid tool for assessing balance and predicting fall risk across various populations, including older adults, individuals with neurological conditions (e.g., stroke, Parkinson's disease), and those recovering from orthopedic surgery. Its high test-retest and inter-rater reliability, as well as its strong construct, criterion, and concurrent validity, support its widespread use in clinical practice and research. However, like any assessment tool, it should be used as part of a comprehensive evaluation that includes other clinical assessments and considerations
Lower Extremity Functional Scale (LEFS) | 11 weeks
  The Lower Extremity Functional Scale (LEFS) is a self-reported questionnaire used by physical therapists and other healthcare providers to assess a person's functional ability related to lower extremity (leg) tasks. It is widely used to evaluate the degree of difficulty experienced by individuals with lower extremity injuries or conditions in performing various daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Saleem, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed IA. The effect of sakiyo training on interactive agility, offensive and defensive foot movements, and their relationship to the level of kata performance. journal of Theories and Applications of physical education sport sciences.2022; 6(1): 2636-3925.